CLINICAL TRIAL: NCT05700357
Title: Comparison of Different Local Anesthetic Volumes of Thoracic Paravertebral Block Application in Post-thoracotomy Analgesia
Brief Title: Different Local Anesthetic Volumes for TPVB in Post-thoracotomy Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nilgün Zengin, Principal İnvestigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-22-3143
Record Dates: First submitted 2023-01-07; First posted 2023-01-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Thoracic Paravertebral Block; Thoracotomy; Postoperative Analgesia; Acute Pain; Local Anesthetic
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracic Paravertebral Block 20 ml (Active Comparator): In patients who are planned to have a thoracic paravertebral block, the needle will be advanced to the paravertebral area with ultrasound-guided in-plane technique. 20 ml of 0.25% bupivacaine will be injected into this area.
  Interventions: Procedure: TPVB with 20 ml
- Thoracic Paravertebral Block 25 ml (Active Comparator): In patients who are planned to have a thoracic paravertebral block, the needle will be advanced to the paravertebral area with ultrasound-guided in-plane technique. 25 ml of 0.25% bupivacaine will be injected into this area.
  Interventions: Procedure: TPVB with 25 ml
- Thoracic Paravertebral Block 30 ml (Active Comparator): In patients who are planned to have a thoracic paravertebral block, the needle will be advanced to the paravertebral area with ultrasound-guided in-plane technique. 30 ml of 0.25% bupivacaine will be injected into this area.
  Interventions: Procedure: TPVB with 30 ml

INTERVENTIONS:
Procedure: TPVB with 20 ml — The thoracic paravertebral block will be applied to the patients with 20 ml of 0.25% bupivacaine under real-time ultrasound guidance.
  Arms: Thoracic Paravertebral Block 20 ml
Procedure: TPVB with 25 ml — The thoracic paravertebral block will be applied to the patients with 25 ml of 0.25% bupivacaine under real-time ultrasound guidance.
  Arms: Thoracic Paravertebral Block 25 ml
Procedure: TPVB with 30 ml — The thoracic paravertebral block will be applied to the patients with 30 ml of 0.25% bupivacaine under real-time ultrasound guidance.
  Arms: Thoracic Paravertebral Block 30 ml

SUMMARY:
Thoracotomy is one of the most painful operations known. Therefore, it causes severe acute pain. If pain is not controlled, it increases the frequency of postoperative pulmonary complications and postoperative morbidity. It can even cause chronic pain in the future. Thoracic epidural analgesia (TEA) is the gold standard method in the treatment of pain after thoracotomy. Thoracic paravertebral block (TPVB) is known as the most effective method after TEA. The fact that TPVB has fewer side effects than TEA increases the use of TPVB. There is no consensus on the dose of analgesia in studies. In the literature, volumes between 20 ml and 30 ml are frequently used for TPVB in recent years. This study, it was aimed to compare the efficacy of 20 ml, 25 ml, and 30 ml volumes of TPVB with local anesthetic at the same concentration (0.25% bupivacaine) on postoperative analgesia in patients undergoing thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* American Society of Anesthesiologists (ASA) physical status I-II-III
* BMI 18 to 40 kg/m2
* Elective thoracotomy surgery

Exclusion Criteria:

* Patient refusing the procedure
* Emergency surgery
* History of chronic opioid or analgesic used

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-11-28 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | 1st hour after surgery
  Pain will be assessed at the first-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 2nd-hour after surgery
  Pain will be assessed at the 2nd-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 4th-hour after surgery
  Pain will be assessed at the 4th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 12th-hour after surgery.
  Pain will be assessed at the 12th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 24th-hour after surgery.
  Pain will be assessed at the 24th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 48th-hour after surgery.
  Pain will be assessed at the 48th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Morphine Consumption | 24 hours after surgery
  Morphine consumption for 24 hours will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No